CLINICAL TRIAL: NCT05099718
Title: Effect of Hyaluronic Acid on Oral Mucosal Wound Healing - Focus on Pain and Re-epithelisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Andreas Stavropoulos, Prof, Malmö University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-01018
Record Dates: First submitted 2021-10-09; First posted 2021-10-29 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Soft Tissue Wound Healing
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyaluronic acid (Experimental): Application 3-times per day for 7 days.
  Interventions: Procedure: palatal soft tissue harvesting; Device: Hyaluronic acid
- Saline solution (Placebo Comparator): Application 3-times per day for 7 days.
  Interventions: Procedure: palatal soft tissue harvesting; Other: Saline solution (placebo)

INTERVENTIONS:
Procedure: palatal soft tissue harvesting — A 6x2mm palatal soft tissue graft will be harvested.
Device: Hyaluronic acid — application 3-times per day for 7 days
  Arms: Hyaluronic acid
Other: Saline solution (placebo) — application 3-times per day for 7 days
  Arms: Saline solution

SUMMARY:
Establishment of a sufficiently wide and thick keratinized gingival/mucosal tissue cuff around teeth/implants is considered of importance for long-term stability. This can more readily be achieved by means of autogenous soft tissue grafts harvested from the palate than with soft tissue substitutes. However, this often implies the creation of an open palatal wound involving secondary intention healing. The aim of this randomized controlled, split-mouth, clinical trial is to assess the effect of a hyaluronic acid containing commercial product on wound healing and patient morbidity after palatal soft tissue harvesting. Altogether, 20 volunteers will be recruited. An individualized splint containing 2 symmetrically located contralateral cylindrical openings will be used for standardized soft tissue harvesting (6 mm in Ø, 2 mm in depth). Soft tissue grafts will be harvested randomly from the right or left side and patients will be monitored for 3 weeks followed by a 1-month wash-out period prior to harvesting the second soft tissue graft from the other side. Participants will randomly start treating the palatal wound either with the test product (GUM Aftaclear Gel, Sunstar Suisse SA, Etoy, Switzerland; 0.3%) or saline solution for 7 days to promote the healing process, which will be reversed for the second round. Patient-related outcomes (morbidity, discomfort, taste alteration, pain killer consumption), frequency of bleeding events, defect closure (area, volume), and microbial colonisation will be recorded and analysed for any differences between the control and test product. Further, in 6 additional volunteers, biopsies of the healing wound are collected in a similar fashion as described above, but with the use of a larger stent in order to harvest also pristine surrounding tissues for histological analysis; biopsies are collected up to 14 days of healing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years,
* systemically healthy,
* healthy periodontal conditions at the experimental region or conditions not interfering with proper biopsy harvesting,
* no known sensitivity to HY,
* no uncontrolled diabetes mellitus,
* no radiotherapy or chemotherapy,
* no current pregnancy or breastfeeding,
* no hormonal diseases,
* no infectious diseases,
* no autoimmune diseases or under immunotherapy,
* no systemic bone disease,
* no wound healing disorders or acute inflammatory/infectious processes,
* no systemic diseases with implications on mucous membranes (e.g., Morbus Crohn),
* no increased risk of bleeding (i.e., patient with coagulation disorders or under anticoagulant therapy, and
* no heavy smokers (i.e., no regular tobacco consumption > 10 cigarettes/day).

Exclusion Criteria:

* not meeting the inclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
pain / discomfort (burning) perception by means of a 100 mm VAS | 3 days
  0 indicates no pain, 100 indicates maximum pain
pain / discomfort (burning) perception by means of a 100 mm VAS | 7 days
  0 indicates no pain, 100 indicates maximum pain
pain / discomfort (burning) perception by means of a 100 mm VAS | 14 days
  0 indicates no pain, 100 indicates maximum pain
pain / discomfort (burning) perception by means of a 100 mm VAS | 21 days
  0 indicates no pain, 100 indicates maximum pain

SECONDARY OUTCOMES:
pain killer consumption | 3 days
  amount of pills taken
pain killer consumption | 7 days
  amount of pills taken
pain killer consumption | 14 days
  amount of pills taken
pain killer consumption | 21 days
  amount of pills taken
disturbance while eating or drinking by means of a 100 mm VAS | 3 days
  0 indicates no disturbance, 100 indicates maximum disturbance
disturbance while eating or drinking by means of a 100 mm VAS | 7 days
  0 indicates no disturbance, 100 indicates maximum disturbance
disturbance while eating or drinking by means of a 100 mm VAS | 14 days
  0 indicates no disturbance, 100 indicates maximum disturbance
disturbance while eating or drinking by means of a 100 mm VAS | 21 days
  0 indicates no disturbance, 100 indicates maximum disturbance
taste alteration experience by means of a 100 mm VAS | 3 days
  0 indicates no alteration, 100 indicates maximum alteration
taste alteration experience by means of a 100 mm VAS | 7 days
  0 indicates no alteration, 100 indicates maximum alteration
taste alteration experience by means of a 100 mm VAS | 14 days
  0 indicates no alteration, 100 indicates maximum alteration
taste alteration experience by means of a 100 mm VAS | 21 days
  0 indicates no alteration, 100 indicates maximum alteration
frequency of re-bleeding | 3 days
  number of events
frequency of re-bleeding | 7 days
  number of events
frequency of re-bleeding | 14 days
  number of events
frequency of re-bleeding | 21 days
  number of events
re-epithelialised defect area (by means of standardized photographs) | 3 days
  mm2
re-epithelialised defect area (by means of standardized photographs) | 7 days
  mm2
re-epithelialised defect area (by means of standardized photographs) | 14 days
  mm2
re-epithelialised defect area (by means of standardized photographs) | 21 days
  mm2
re-epithelisation by colorimetric digital assessment of the calibrated photographs | 3 days
  colorimetric assessment
re-epithelisation by colorimetric digital assessment of the calibrated photographs | 7 days
  colorimetric assessment
re-epithelisation by colorimetric digital assessment of the calibrated photographs | 14 days
  colorimetric assessment
re-epithelisation by colorimetric digital assessment of the calibrated photographs | 21 days
  colorimetric assessment
changes in total and specific bacterial counts | 3 days
  log values
changes in total and specific bacterial counts | 7 days
  log values
changes in total and specific bacterial counts | 14 days
  log values
defect volume fill by overlay of the intraoral scans | 3 days
  mm3
defect volume fill by overlay of the intraoral scans | 7 days
  mm3
defect volume fill by overlay of the intraoral scans | 14 days
  mm3
defect volume fill by overlay of the intraoral scans | 21 days
  mm3
food restrictions (yes/no) | 3 days
food restrictions (yes/no) | 7 days
food restrictions (yes/no) | 14 days
food restrictions (yes/no) | 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Odontology, Malmo University, Malmo, Sweden